CLINICAL TRIAL: NCT03032029
Title: Registry on the Treatment of Central and Complex Sleep-Disordered Breathing With Adaptive Servo-Ventilation
Acronym: READ-ASV
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Collaborators: CRI-The Clinical Research Institute GmbH (Industry); University Hospital Regensburg (Other)
Responsible Party: Sponsor
Other Study IDs: READ-ASV_Reg_Protoc_170404; Protocol 2019-04-16 (Other: ResMed); NCT04331821 (obsolete NCT alias)
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-01

CONDITIONS: Central Sleep Apnea; Complex Sleep Apnea; Obstructive Sleep Apnea; Mixed Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Central; Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Adaptive Servo-Ventilation — Adaptive Bi-Level positive airway pressure with a targeted minute ventilation and auto-adjusting expiratory pressure level.

SUMMARY:
Phase 1: The European ASV Registry (short name) will investigate the use of Adaptive Servo-Ventilation in non-heart failure conditions. The purpose is to examine the effects of ASV on quality of life, daytime symptoms and sleep, to describe usage patterns of ASV with regards to patient characteristics and to document adverse events related to therapy for a therapy safety analysis. A pilot phase will enrol at least 200 patients to test the feasibility of the registry. After the pilot phase will be completed and an intermediate data analysis had been performed, the registry will be expanded over several countries across Europe with the goal of enrolling up to 800 patients over a period of 5 years. Phase 2: The READ-ASV Registry (short name) will investigate the use of Adaptive Servo-Ventilation in non-heart failure conditions. The purpose is to examine the effects of ASV on quality of life, daytime symptoms and sleep, to describe usage patterns of ASV with regards to patient characteristics and to document adverse events related to therapy for a therapy safety analysis.

DETAILED DESCRIPTION:
Phase 1: The collection of data will be performed during the course of clinical routine. In regular clinical practice, a first control visit (i.e. Follow-up number one) should occur during the first 6 months. Further follow-up visits are only indicated when the patient is reporting problems during the course of therapy. We recommend FU visit at least once year (after the first routine FU visit). Each patient will be included for 6 months, the total duration of phase 1 of the registry. Phase 2: The pilot phase 1 enrolled over 200 patients. After completion of the pilot phase the registry expands to 1 additional country in Europe with the goal of enrolling up to 800 patients over a period of 4 years. The collection of data will be performed during the course of clinical routine. In regular clinical practice, a first control visit (i.e. Follow-up number one) should occur after the first 12 months of therapy use. Further follow-up visits are only indicated when the patient is reporting problems during the course of therapy. Each patient will be included for a maximum of 15 months, whereas serious events will be tracked throughout the total duration of phase I and II of the registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients over ≥18 years of Age
* Prescription of ResMed AirCurve 10 CS PaceWave or S9 AutoSet CS PaceWave for treatment of ASV
* Naive to ASV Treatment
* Able to fully understand information on data protection and provide written informed consent

Exclusion Criteria:

- Heart Failure (HF) with a Left Ventricular Ejection Fraction (LVEF) <45% and CSA >50% central apneas of all apneas

Phase 2: Inclusion Criteria:

* ≥ 18 years old.
* Indication for treatment with ASV according to applicable medical guidelines.
* Use of eligible ResMed devices for treatment with ASV according to the Instructions For Use of the corresponding device.
* Naive to ASV treatment (max. 7 days between start of ASV therapy and enrolment).
* Able to fully understand information on data protection and provide written informed consent for use of their medical data.

Phase 2: Exclusion Criteria:

* Chronic, symptomatic heart failure (NYHA 2-4) with reduced left ventricular ejection fraction (LVEF ≤ 45%) and moderate to severe predominant central sleep apnea.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry shall include adult individuals with a prescription of ASV therapy. Indications are sleep-related breathing disorders, including obstructive, central or complex sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 847 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life, assessed with the Functional Outcomes of Sleep Questionnaire (FOSQ) by comparing the score at baseline with the 12 months follow-up. | 12 months
  The Functional Outcomes of Sleep Questionnaire had been developed to comprehensively capture the impact of sleeping disorders in relevant daily activities as for instance general activity, vigilance, intimacy, fitness and social life.
Phase 2: Quality of Life, assessed with the Functional Outcomes of Sleep Questionnaire (FOSQ) by comparing the score at baseline with the follow-up after 12 months. | Baseline to 12 months
  The Functional Outcomes of Sleep Questionnaire had been developed to comprehensively capture the impact of sleeping disorders in relevant daily activities as for instance general activity, vigilance, intimacy, fitness and social life. The FOSQ consists of 30 questions, answer options ranging from 4 (no problems) to 1(severe problems) or 0(not applicable) adding up to a total score between 5(worst functional status)-20(best functional status).

SECONDARY OUTCOMES:
Daytime symptoms assessed with the EuroQoL (EQ-5D) by comparing the answers at baseline with answers at the follow-up at 12 months. | 12 months
  The EQ-5D is a standardized questionnaire used to measure the health of patients. It is applicable in a large number of conditions and treatments and provides a simple descriptive profile and a single index value to define a state of health (mobility, self-care ability, activities, discomfort, anxiety).
Daytime sleepiness assessed with the Epworth Sleepiness Scale (ESS) by comparing the score at baseline with the follow-up after 12 months. | 12 months
  The Epworth or Epworth Sleepiness Scale questionnaire assesses excessive daytime sleepiness. It determines the probability of falling asleep in the context of 8 common situations in daily life. The patient self assesses, on a level of 0 to 3, drowsiness over the past few weeks. The maximum total score is 24.
Quality of Sleep assessed with the Pittsburgh Sleep Quality Index (PSQI) at baseline compared with the follow-up after 12 months. | 12 months
  The PSQI includes 19 self-assessment questions and 5 questions asked to the spouse or roommate (if any).The 19 self-assessment questions combine to give 7 components of the overall score, with each component receiving a score of 0-3.
  A score of 0 indicates that there is no difficulty while a score of 3 indicates the existence of severe difficulties. The 7 components of the score add up to give an overall score ranging from 0 to 21 points, 0 meaning that there is no difficulty, and 21 indicating difficulties.
Therapy compliance assessed by the hours of usage per night. | 6 months
  Usually, compliance is defined as device usage of ˃4h/night in ˃70% of nights to see effects on the Status of health. However, a usage of ≥ 3 hours might improve a patient's outcome: Data on úsage of ASV and outcomes is scarce. Since the aim of the study is to assess compliance, the data of the device has to be carefully analysed in connection with the outcomes.
Apnea-Hypopnea-Index assessed by the number of Apneas and hypopneas per hour. | 6 months
  The number of apneas and hypopneas per hour will be counted during the total time of sleep of a Patient, added up and divided by the hours of sleep. The result is an index, which indicates mild sleep apnea (AHI between 5-15 Events/hour), moderate sleep apnea (15-30 Events per hour) or severe sleep apnea (more than 30 Events per hour).
Central Apnea Index assessed by the number of central apneas per hour. | 6 months
  The number of central apneas - where the respiratory effort stops - per hour will be counted during the total time of sleep of a patient, added up and divided by the hours of sleep. The result is an index, which indicates mild central sleep apnea (AHI below 5 Events/hour), moderate central sleep apnea (5-15 Events per hour) or severe central sleep apnea (more than 15 Events per hour).
Safety of ASV therapy assessed by documenting the number of adverse Events and the number of hospitalizations at the Overall end of the study. | 6 months
  Adverse Events of Special Interest (e.g. Skin irritation or wound, Skin rashes, Conjunctivitis, Dryness of the upper airways, Therapy intolerance (pressure), Mask issues, leaks,Technical problems of the device) will be document as well as the number of Hospital stays during the study period.
Phase 2: Daytime symptoms assessed with the EuroQoL (EQ-5D) by comparing the answers at baseline with answers at the follow-up at 12 months. | Baseline to 12 months
  The EuroQoL-5Dimension is a standardized questionnaire used to measure the health of patients. It is applicable in a large number of conditions and treatments. It defines 5 health-states: mobility, self-care ability, activities, discomfort, anxiety. The states of health will be described by rating them from 1(no problems) to 5 (extreme problems). The outcomes can either be displayed as mean (+/-SD) or percentages of patients rating their health state with a certain score. The combined 5 heath-states rating (e.g.11111, 12345 etc.) may be converted to a single index value (index value calculator must be ordered from the manufacturer. The EQ-5D comprises a visual analogue scale ranging from 0=worst health to 100=best health.
Phase 2: Daytime sleepiness assessed with the Epworth Sleepiness Scale (ESS) by comparing the score at baseline with the follow-up after 12 months. | Baseline to 12 months
  The Epworth or Epworth Sleepiness Scale questionnaire assesses excessive daytime sleepiness. It determines the probability of falling asleep in the context of 8 common situations in daily life. The patient self-assesses, on a level of 0 to 3, drowsiness over the past few weeks. The maximum total score is 24 (worst level of daytime sleepiness).
Phase 2: Therapy compliance assessed by the hours of usage per night. | Baseline to 12 months
  Usually, compliance is defined as device usage of ˃4h/night in ˃70% of nights to see effects on the Status of health. However, a usage of ≥ 3 hours might improve a patient's outcome: Data on usage of ASV and outcomes is scarce. Since the aim of the study is to assess compliance, the data of the device has to be carefully analyzed in connection with the outcomes.
Phase 2: Rate of hospitalizations for cardiovascular or respiratory cause per year of follow-up. | 12 months
  All unplanned hospitalizations will be recorded as serious adverse events and assessed for cause of hospitalisation: cardiovascular or respiratory cause.
Phase 2: Rate of all-cause deaths per year of follow-up. | 12 months
  All deaths will be recorded. Cause of death will be assessed through the documentation in the study centers.

CONTACTS AND LOCATIONS:
Locations (29):
- Denmark (2):
  - Sjællands Universitetshospital/Zealand University Hospital Køge, Køge
  - Odense Universitetshospital, Odense
- Centre Hospitalier Universitaire Grenoble Alpes, Grenoble, France
- Germany (19):
  - Schlaf- und Beatmungszentrum, Blaubeuren Abbey, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - Klinik für Pneumologie, Schlaf- und Beatmungsmedizin, Kempten (Allgäu), Bavaria
  - Klinikum Landshut, Landshut, Bavaria
  - Klinikum Nürnberg-Med Klinik 3, Nuremberg, Bavaria
  - University Hospital Regensburg, Regensburg, Bavaria
  - Medizinisches Zentrum, Bad Lippspringe, North Rhine-Westphalia
  - Praxis für Lunge, Herz und Schlaf, Bielefeld, North Rhine-Westphalia
  - Christophorus Kliniken, Dülmen, North Rhine-Westphalia
  - Klinik für Schlafmedizin Düsseldorf Grand Arc, Düsseldorf, North Rhine-Westphalia
  - Ruhrlandklinik Essen, Essen, North Rhine-Westphalia
  - Lungenklinik Hemer, Hemer, North Rhine-Westphalia
  - Evangelisches Krankenhaus Herne, Herne, North Rhine-Westphalia
  - Praxis für Pneumologie, Allergologie, Schlafmedizin Dr. med Christoph Stolpe, Ibbenbueren, North Rhine-Westphalia
  - Fachkrankenhaus Kloster Grafschaft, Schmallenberg, North Rhine-Westphalia
  - Marienkrankenhaus Soest, Soest, North Rhine-Westphalia
  - ZMS Zentrum für medizinische Studien, Warendorf, North Rhine-Westphalia
  - Universitätsklinikum SH, Lübeck, Schleswig-Holstein
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Hospital Sao Joao, Porto
- Spain (3):
  - Hospital de Cruces, Barakaldo
  - Hospital Clinic, Barcelona
  - Hospital General de Asturias, Oviedo
- Switzerland (2):
  - Inselspital, Bern
  - Centre d' investigation et de recherche sur le sommeil, Lausanne

REFERENCES:
- [Background] Arzt M, Munt O, Pepin JL, Heinzer R, Kubeck R, von Hehn U, Ehrsam-Tosi D, Benjafield A, Woehrle H. Registry on the Treatment of Central and Complex Sleep-Disordered Breathing with Adaptive Servo-Ventilation (READ-ASV): protocol and cohort profile. ERJ Open Res. 2023 Apr 17;9(2):00618-2022. doi: 10.1183/23120541.00618-2022. eCollection 2023 Mar. PMID 37077553
- [Background] Arzt M, Munt O, Pepin JL, Heinzer R, Kubeck R, von Hehn U, Ehrsam-Tosi D, Benjafield AV, Woehrle H. Effects of Adaptive Servo-Ventilation on Quality of Life: The READ-ASV Registry. Ann Am Thorac Soc. 2024 Apr;21(4):651-657. doi: 10.1513/AnnalsATS.202310-908OC. PMID 38241012
- [Derived] Arzt M, Munt O, Kuebeck R, Woehrle H, Heinzer R, Benjafield AV, Pepin JL. Adaptive Servo-Ventilation for Treatment-Emergent Central Sleep Apnea: The READ-ASV Registry. Ann Am Thorac Soc. 2025 Oct;22(10):1546-1553. doi: 10.1513/AnnalsATS.202502-210OC. PMID 40359269
- [Derived] Pepin JL, Benjafield AV, Munt O, Woehrle H, Heinzer R, Arzt M; READ-ASV Investigators. Treatment of sleep-disordered breathing in opioid users with adaptive servo-ventilation: a subgroup analysis of the European READ-ASV registry. J Clin Sleep Med. 2025 Jul 1;21(7):1227-1232. doi: 10.5664/jcsm.11652. PMID 40135691